CLINICAL TRIAL: NCT00565955
Title: Effect Of Addition of Oral Montelukast to Standard Treatment in Acute Moderate to Severe Asthma in Children Between 5-15 Years of Age - A Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Effect of Addition of Oral Montelukast to Standard Treatment in Acute Moderate to Severe Asthma in Children
Acronym: Montelukast
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: VIVEK KUMAR TODI, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: vivek
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Bronchial Asthma
Keywords: Montelukast; Acute Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A1 (Active Comparator): Children Between 5-15 Years of Age Receiving Montelukast
  Interventions: Drug: montelukast
- A2 (Placebo Comparator): Children Between 5-15 Years of Age Receiving Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: montelukast — Standard case management will be carried out as per guidelines given by British Thoracic Society. All patients will receive montelukast or similar looking placebo tablets. The doses of montelukast will be as follows:
  5-12 years: 5 mg chewable tablet of montelukast; > 12 years: 10 mg chewable tablet of montelukast. Study drug will be administered at time of administration of steroid.
  Arms: A1
Drug: Placebo — The patients will receive placebo tablets.
  Arms: A2

SUMMARY:
Available evidences show a role of oral montelukast in acute asthma. Safety of oral montelukast is well established in children, as evidenced by use of oral montelukast in long term management of asthma.

Therefore, the investigators planned this study to see the effect of oral montelukast as add on therapy to standard treatment in acute moderate to severe asthma in children between 5-15 years of age.

HYPOTHESIS:

Addition of single dose of oral montelukast to standard therapy in acute moderate to severe asthma in children aged 5-15 years will reduce the modified pulmonary index score to less than 9 in 90% children compared to 70% in children receiving a placebo.

DETAILED DESCRIPTION:
Leukotrienes plays an important role as mediator for inflammatory changes in acute as well as chronic asthma. There are three randomized controlled trials involving 274 adult patients with acute asthma who were treated with montelukast (intravenous in 2 and intravenous and oral in one study) to see the beneficial response in spirometry. All the studies showed significant improvement in FEV1 in first 2 hours. These studies show that oral montelukast causes improved pulmonary function and has a rapid onset of action. However, these studies are carried out in adults. Safety of oral montelukast is well established in children, as evidenced by use of oral montelukast in long term management of asthma.

Therefore, we planned this study to see the effect of oral montelukast as add on therapy to standard treatment in acute moderate to severe asthma in children between 5-15 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-15 years of age, either sex seeking treatment with acute moderate to severe asthma in pediatric casualty/ chest clinic/ out patient services. Acute moderate to severe asthma is defined as modified pulmonary index score of more than 9.

Exclusion Criteria:

* Children with life threatening asthma (poor respiratory efforts, cyanosis, altered sensorium).
* Children who had received montelukast within one week of arrival.
* Children with other chronic respiratory conditions (including congenital lung abnormalities) like tuberculosis, cystic fibrosis or other acute illnesses that would complicate current treatment and response for asthma.
* Children with altered sensorium/unable to take oral medication.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Reduction in modified pulmonary index score (MPIS) to less than 9 at the end of 4 hours. | 4 hours

SECONDARY OUTCOMES:
Change in FEV1 at the end of 4 hours | 4 hours
Adverse effects: Headache, nausea, vomiting, abdominal pain | 4 hours
Need for hospitalization | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: SUSHIL K KABRA, Study Director — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Todi VK, Lodha R, Kabra SK. Effect of addition of single dose of oral montelukast to standard treatment in acute moderate to severe asthma in children between 5 and 15 years of age: a randomised, double-blind, placebo controlled trial. Arch Dis Child. 2010 Jul;95(7):540-3. doi: 10.1136/adc.2009.168567. Epub 2010 Jun 3. PMID 20522464